CLINICAL TRIAL: NCT00138658
Title: A Phase 1-2 Study of Weekly OGX-011 Plus a Gemcitabine/Platinum-Based Regimen in Patients With Stage IIIB or IV Non Small Cell Lung Cancer
Brief Title: A Study of OGX-011/Gemcitabine/Platinum-Based Regimen in Stage IIIB/IV Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OGX-011-05
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Results first posted 2012-01-10 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; custirsen sodium; OGX-011; Stage IIIB or IV advanced non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — OGX-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: custirsen sodium — Custirsen sodium (OGX-011) was to be infused intravenously over 2 hours on Days -7, -5, and 3 of Cycle 1 (pretreatment loading dose). OGX 011 was then to be infused for 2 hours weekly on Days 1, 8, and 15 of a 21-day cycle. Gemcitabine (GEM) was to be infused intravenously for 30 minutes on Days 1 and 8 and either cisplatin (CIS) or carboplatin (CARBO) were to be infused intravenously on Day 1 of this 21-day cycle. Patients were to receive a maximum of 6 cycles (1 cycle = 21 days)
  Other Names: OGX-011; TV-1011

SUMMARY:
This clinical study will help determine if giving OGX-011 (custirsen sodium) in combination with gemcitabine (GEM) and cisplatin (CIS) or carboplatin (CARB) is a safe and effective treatment for patients with lung cancer. This study will help to assess the safety and anti-tumor effect of OGX-011 when given to patients in combination with GEM and CIS/CARB.

DETAILED DESCRIPTION:
OGX-011 is an experimental drug that has been shown to increase the effectiveness of commonly used cancer therapies such as chemotherapy, radiation and hormone therapy in several kinds of cancer types in animals. OGX-011 is being studied in the treatment of cancer patients in combination with chemotherapy. In humans, OGX-011 in combination with hormone therapy has been shown to decrease the tissue levels of a protein called clusterin, which can be overproduced in cancer cells. Clusterin has been found to block cell death and makes cells more resistant to cancer therapy. Gemcitabine (GEM), cisplatin (CIS) and carboplatin (CARB) have been approved by Health Canada and the Food and Drug Administration in the United States for the treatment of patients with lung cancer.

OGX-011 was administered as a 2-hr intravenous (IV) infusion on Days -7, -5, and -3 prior to Cycle 1, then weekly on Days 1, 8, 15 of each 21-day cycle; GEM was infused IV after OGX-011 on Days 1 and 8; either CIS or CARB was infused IV after GEM on Day 1 of each cycle. Six cycles of treatment were planned. Most patients received OGX-011 at 640 mg, but 3 patients received OGX-011 at 480 mg dose; OGX-011 dose groups were combined due to the small number of patients who received 480 mg.

ELIGIBILITY:
Inclusion Criteria

1. Patients must have a histologically or cytologically confirmed diagnosis of NSCLC and must not have had chemotherapy or biological therapy for their disease.
2. Stage IIIB (N3 and/or pleural or pericardial effusion) or IV disease that is not amenable to either surgery or radiation therapy of curative intent.
3. Life expectancy of ≥ 12 weeks
4. If patient has had prior radiation therapy: lesion(s) used for determination of response was not previously irradiated or has increased in size since the completion of radiotherapy; and patient has recovered from any toxicity from the radiotherapy.
5. Radiotherapy to lesion(s) used for determination of response was completed at least 6 weeks prior to treatment; radiotherapy to other sites was completed at least 2 weeks prior to treatment.
6. At least one unidimensionally measurable lesion meeting Response Evaluation Criteria in Solid Tumors [RECIST] (at least 10 mm in longest diameter by spiral computed tomography [CT] scan, or at least 20 mm by standard techniques).
7. ECOG status must be ≤ 1

Exclusion Criteria

1. Prior chemotherapy or biological therapy (approved or experimental) for NSCLC, including adjuvant and neoadjuvant treatment.
2. Presence of central nervous system (CNS) metastases, unless the patient has completed successful local therapy for CNS metastases, with the exception of leptomeningeal disease for which patients will be excluded. Patients must be off corticosteroids for at least 21 days prior to starting treatment.
3. Second primary malignancy (except in situ carcinoma of the cervix, adequately treated non-melanomatous skin cancers, clinically localized prostate cancer, superficial bladder cancer or other malignancy treated at least 3 years previously with no evidence of recurrence).
4. Patients eligible for combined modality therapy with curative intent as defined by the combination of chemotherapy, radiation therapy and/or surgery. (This criteria is intended to exclude patients with stage IIIB disease, as defined by the presence of N3 nodal status, who have been reported to have cure rates as high as 10% when treated with combined modality therapy.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2004-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janessa Laskin, M.D., Principal Investigator — BCCA, Vancouver Clinic
Locations (15):
- United States (6):
  - LAC-USC Medical Center, Los Angeles, California
  - University of Southern California Norris, Los Angeles, California
  - New York Oncology Hematology, Albany, New York
  - Oregon Health and Science University, Portland, Oregon
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Mary Crowley Medical Research Center, Dallas, Texas
- Canada (9):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BC Cancer Agency, Fraser Valley Centre, Surrey, British Columbia
  - BC Cancer Agency, Vancouver Center, Vancouver, British Columbia
  - Dr. H. Bliss Murphy Cancer Center, St. John's, Newfoundland and Labrador
  - Royal Victoria Hospital of Barrie, Barrie, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Toronto Sunnybrook Regional Cancer Center, Toronto, Ontario
  - Hopital Laval, Ste-Foy, Quebec

REFERENCES:
- [Result] Laskin JJ, Nicholas G, Lee C, Gitlitz B, Vincent M, Cormier Y, Stephenson J, Ung Y, Sanborn R, Pressnail B, Nugent F, Nemunaitis J, Gleave ME, Murray N, Hao D. Phase I/II trial of custirsen (OGX-011), an inhibitor of clusterin, in combination with a gemcitabine and platinum regimen in patients with previously untreated advanced non-small cell lung cancer. J Thorac Oncol. 2012 Mar;7(3):579-86. doi: 10.1097/JTO.0b013e31823f459c. PMID 22198426

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 15 institutions with a primary focus on oncology and located in the United States and Canada. The date of the first screening visit was November 2004 and the last survival followup was February 2010.
Pre-assignment Details: Four subjects who were assigned a study ID number were determined to be ineligible (i.e., failed one or more inclusion/exclusion criteria) and were never treated.
Groups:
- OGX-011 - Intent to Treat Analysis Set: Custirsen sodium (OGX-011) was to be infused intravenously over 2 hours on Days -7, -5, and -3 of Cycle 1 (Pretreatment loading doses). OGX-011 was then to be infused for 2 hours weekly on Days 1, 8, and 15 of a 21-day cycle. Gemcitabine (GEM) was to be infused IV for 30 minutes on Days 1 and 8 and either cisplatin (CIS) or carboplatin (CARBO) were to be infused IV on Day of the 21-day cycle. Patients were to receive a maximum of 6 cycles (1 cycle =21 days). Most patients received OGX-011 at 640 mg; but 3 patients received a 480 mg dose. The 2 dose groups were combined due to the small number of patients who received 480 mg. All patients who received at least one dose of OGX-011 were included in the Intent to Treat Analysis Set.
Period: Overall Study
Arm/Group | OGX-011 - Intent to Treat Analysis Set
Started | 81
Completed | 20
Not Completed | 61
Not completed — Adverse Event | 23
Not completed — Death | 1
Not completed — Disease Progression | 21
Not completed — Physician Decision | 11
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | OGX-011 - Intent to Treat Analysis Set
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 25
Age Continuous [Mean (Full Range); unit: years] | 60.4 [43 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 72
  More than one race | 0
  Unknown or Not Reported | 1
Baseline ECOG [Number; unit: participants] — The ECOG score is a performance status which attempts to quantify cancer patients' general well-being.
  Grade 0=Fully active, able to carry on all pre-disease performance without restriction.
  Grade 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Grade 2=Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours.
  participants
    ECOG O | 26
    ECOG 1 | 54
    ECOG 2 | 1
Cancer Stage [Number; unit: participants] — Patients enrolled in this study were required to be either Stage IIIB or Stage IV.
  Stage IIIB lung cancer is defined as a tumor of any size that has spread to distant lymph nodes, has invaded other structures in the chest (such as the heart or esophagus), or has a malignant pleural effusion (fluid build-up containing cancer cells between the layers lining the lungs).
  Stage IV non-small cell lung cancer is defined as a tumor of any size that has spread (metastasized) to another region of the body or to another lobe of the lungs.
  participants
    Stage IIIB | 15
    Stage IV | 66

OUTCOME MEASURES:

1. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as time from first treatment with OGX-011 to documented evidence of disease progression or date of death. For subjects without disease progression based on RECIST who initiated subsequent anti-cancer therapy, date of progression was defined as date of initiating new cancer treatment. PFS was censored as of the date of first OGX-011 dose for subjects who failed to return for assessments after screening. For subjects who were still alive and without progressive disease at the time of data cut-off, PFS was censored at date of last disease assessment.
Time Frame: All subjects were followed for a minimum of 3 years after the first dose of OGX-011 or until death.
Population: Number of patients who progressed or died (n=75); data for 6 patients were censored. (PFS was censored at the date of the first dose of OGX-011 for subjects who failed to return for any disease assessments after screening.)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | OGX-011 - Intent to Treat Analysis Set
Number analyzed (Participants) | 75
months | 4.3 [3.0 to 5.3]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as time from date of first treatment with OGX-011 to the date of death from any cause. Overall survival was censored at date of last contact for subjects who were still alive at end of study.
Time Frame: All subjects were followed for a minimum of 3 years after the first dose of OGX-011 or until death.
Population: Number of subjects who died (n=70); n=11 subjects were censored at end of study (10 were alive and 1 was lost to follow up)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | OGX-011 - Intent to Treat Analysis Set
Number analyzed (Participants) | 70
months | 14.1 [9.4 to 17.5]

3. Secondary Outcome: Effect of OGX-011 on Serum Clusterin Levels
Description: To measure the effect of OGX-011 on serum clusterin levels. The drug substance, OGX-011, is an antisense product designed to bind to clusterin mRNA, resulting in the inhibition of the production of human clusterin protein. Therefore, serum clusterin levels were expected to decrease.
Time Frame: Blood samples were collected at baseline and prior to infusion on Cycle 2 Day 1 and Cycle 3 Day 1
Population: 55 evaluable subjects had baseline value and at least one post-baseline serum clusterin assessment.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Mean Reduction in Serum Clusterin From Baseline: The mean reduction in serum clusterin was calculated by determining the difference from baseline to the minimum post baseline level. The reduction in serum clusterin was determined for all subjects who had baseline and at least one post-baseline serum clusterin assessment (n=55).
Arm/Group | Mean Reduction in Serum Clusterin From Baseline
Number analyzed (Participants) | 55
µg/mL | -25.5 (23.1)

4. Secondary Outcome: Cmax of OGX-011
Description: Cmax is a plasma pharmacokinetic parameter that is defined as the maximum observed concentration of drug substance in plasma.
Time Frame: Blood samples were collected as follows. Cycle 1; Day 1: pre-dose, 2 h (EOI), 0.5 h, 1 hr, 1.5 h, 2.5 h, 4 h, 6.5 h and 23.5 h post end of OGX-011 infusion, Day 22: pre-dose Cycle 2.
Population: Data are reported for the 6 subjects who received 640 mg OGX-011. This is the dose to be used in additional Phase 3 studies of OGX-011
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Patients in Phase I Receiving 640 mg of OGX-011: Per protocol, ten subjects enrolled in the Phase I portion of the study. Three subjects received 480 mg; 6 subjects received 640 mg doses of OGX-011; and 1 patient discontinued prior to Cycle 1 Day 1 due to disease progression.
Arm/Group | Patients in Phase I Receiving 640 mg of OGX-011
Number analyzed (Participants) | 6
ng/mL | 64086 (8756)

5. Primary Outcome: Objective Response Rate of OGX-011 in Combination With Gemcitabine/Platinum-based Regimen
Description: Per RECIST Criteria V 1.0 and based on radiographic evaluations a subject was defined as having an objective response (OR) if the subject achieved either a confirmed partial response (PR) or confirmed complete response (CR).
  The evaluations were conducted after every two cycles of treatment for a maximum of 6 cycles.
  CR: disappearance of clinical/radiological evidence of tumor.
  PR: >= 30% decrease in the sum of the longest diameter of target lesions.
  SD: did not fulfill the criteria for CR or PR but not progressive disease.
Time Frame: Based on assessments at baseline and after Cycles 2, 4, and 6. All subjects were followed for survival for a minimum of 3 years after the first dose of OGX-011 or until death.
Population: The efficacy analysis included all 81 subjects that received at least one dose of OGX-011. Of the 25 subjects with CR or PR, 21 subjects had a confirmed response. The other 4 patients did not have confirmatory scans (n=3) or discontinued treatment (N=1).
Measure: Number; unit: percentage of participants
Arm/Group | OGX-011 - Intent to Treat Analysis Set
Number analyzed (Participants) | 81
percentage of participants | 26

6. Secondary Outcome: t1/2 of OGX-011
Description: Plasma half life of OGX-011
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Patients in Phase I Receiving 640 mg of OGX-011
Number analyzed (Participants) | 6
hours | 3.7 (0.43)

7. Secondary Outcome: AUC-0-last
Description: AUC-0-last is the area under the plasma concentration time curve from time 0 to the last last time point (23.5 hrs)
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Patients in Phase I Receiving 640 mg of OGX-011
Number analyzed (Participants) | 6
ng*h/mL | 260747 (42578)

ADVERSE EVENTS:
Time Frame: Displays of adverse events include treatment-emergent events in all subjects who had at least one adverse event with onset on or after the date of administration of the first dose of study treatment through 30 days after the last dose of study treatment.
Description: Adverse events are systematically assessed through regular investigator assessment and laboratory testing that is clearly defined in the protocol.
Arm/Group | OGX-011 - Intent to Treat Analysis Set
Serious Adverse Events (participants affected / at risk) | 32/81
Other Adverse Events (participants affected / at risk) | 81/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OGX-011 - Intent to Treat Analysis Set (N=81)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Chills (General disorders) | 2
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 2
Fatigue (General disorders) | 1
Pain (General disorders) | 1
Bacteraemia (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Cerebrovascular accident (Nervous system disorders) | 3
Ataxia (Nervous system disorders) | 1
Motor dysfunction (Nervous system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Ventricular hypokinesia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Gastric perforation (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Confusional state (Psychiatric disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1
Blindness cortical (Eye disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OGX-011 - Intent to Treat Analysis Set (N=81)
Anaemia (Blood and lymphatic system disorders) | 36
Neutropenia (Blood and lymphatic system disorders) | 36
Thrombocytopenia (Blood and lymphatic system disorders) | 25
Leukopenia (Blood and lymphatic system disorders) | 9
Nausea (Gastrointestinal disorders) | 60
Vomiting (Gastrointestinal disorders) | 48
Fatigue (General disorders) | 57
Chills (General disorders) | 51
Pyrexia (General disorders) | 50
Oedema Peripheral (General disorders) | 25
Chest Pain (General disorders) | 16
Pain (General disorders) | 15
Asthenia (General disorders) | 14
Influenza Like Illness (General disorders) | 7
Chest Discomfort (General disorders) | 6
Constipation (Gastrointestinal disorders) | 47
Diarrhoea (Gastrointestinal disorders) | 28
Abdominal Pain (Gastrointestinal disorders) | 11
Stomatitis (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 9
Abdominal Distension (Gastrointestinal disorders) | 8
Dry Mouth (Gastrointestinal disorders) | 6
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 4
Decreased Appetite (Metabolism and nutrition disorders) | 43
Hypokalaemia (Metabolism and nutrition disorders) | 18
Hypomagnesaemia (Metabolism and nutrition disorders) | 17
Dehydration (Metabolism and nutrition disorders) | 10
Hyponatraemia (Metabolism and nutrition disorders) | 8
Dysgeusia (Nervous system disorders) | 30
Headache (Nervous system disorders) | 29
Dizziness (Nervous system disorders) | 24
Peripheral Sensory Neuropathy (Nervous system disorders) | 8
Paraesthesia (Nervous system disorders) | 7
Hypoaesthesia (Nervous system disorders) | 5
Tremor (Nervous system disorders) | 5
Neuropathy Peripheral (Nervous system disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33
Cough (Respiratory, thoracic and mediastinal disorders) | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 28
Rash (Skin and subcutaneous tissue disorders) | 21
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 11
Urticaria (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 17
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 14
Back Pain (Musculoskeletal and connective tissue disorders) | 12
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 9
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 5
Neck Pain (Musculoskeletal and connective tissue disorders) | 4
Weight Decreased (Investigations) | 14
Blood Creatinine Increased (Investigations) | 13
Creatinine Renal Clearance Decreased (Investigations) | 11
Alanine Aminotransferase Increased (Investigations) | 10
Blood Alkaline Phosphatase Increased (Investigations) | 10
Aspartate Aminotransferase Increased (Investigations) | 9
Haemoglobin Decreased (Investigations) | 8
Platelet Count Decreased (Investigations) | 6
Insomnia (Psychiatric disorders) | 27
Anxiety (Psychiatric disorders) | 17
Confusional State (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 5
Oral Candidiasis (Infections and infestations) | 8
Oral Herpes (Infections and infestations) | 4
Urinary Tract Infection (Infections and infestations) | 4
Phlebitis (Vascular disorders) | 8
Hypotension (Vascular disorders) | 5
Flushing (Vascular disorders) | 5
Hot Flush (Vascular disorders) | 5
Hypertension (Vascular disorders) | 5
Tinnitus (Ear and labyrinth disorders) | 15
Contusion (Injury, poisoning and procedural complications) | 7
Vision Blurred (Eye disorders) | 4
Tachycardia (Cardiac disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review proposed written or oral material which describes the results of the Study prior to public release and can embargo communications for a period that is less than or equal to 60 days from the time submitted to the sponsor for review.

The results from one institution shall not be presented before the multi-center publication. If there is no multi-center publication within 12 months after the Study completion the Investigator shall have the right to publish the results.